CLINICAL TRIAL: NCT00802009
Title: Dexamethasone and Analgesic Duration After Supraclavicular Brachial Plexus Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Richard Brull, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-0896-B
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Anesthesia
Keywords: ultrasound-guided regional anesthesia; nerve block; brachial plexus; mepivicaine; dexamethasone; hand wrist surgery; duration; anesthetic duration following brachial plexus/nerve block for hand/wrist surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dexamethasone 8mg added to routine local anesthetic during brachial plexus blockade.
  Interventions: Drug: Dexamethasone; Drug: Mepivicaine
- 2 (Active Comparator): Routine anesthetic solution (30 cc 1.5% mepivicaine) used during brachial plexus blockade.
  Interventions: Drug: Mepivicaine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8 milligrams (liquid) will be added to standard anesthetic solution administered during routine brachial plexus nerve blockade.
  Arms: 1
Drug: Mepivicaine — Standard anesthetic solution administered during routine brachial plexus nerve blockade.

SUMMARY:
Patients undergoing surgery of the hand often are treated with a nerve block in the shoulder/neck area that provides anesthesia/numbing during surgery. Nerve blocks usually last for a few hours after surgery and provide pain relief for this period. It may be possible to extend the duration of anesthesia by using a steroid, which has anti-inflammtory properties. This study will compare the duration of the nerve block when dexamethasone (steroid) is added to the anesthetic injected around the nerve.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having unilateral hand or forearm surgery under Supraclavicular brachial plexus blockade.
2. ASA I-III
3. Age 18-60
4. BMI < 35

Exclusion Criteria:

1. Patients with a known history of hypersensitivity to local anesthetics and dexamethasone.
2. Contra-indication to regional anesthesia/ supraclavicular brachial plexus blockade e.g. bleeding diathesis, coagulopathy.
3. Peripheral neuropathy.
4. Peptic ulcer disease.
5. Diabetes Mellitus.
6. Inability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Duration of anesthesia | hourly for first 24 hours; daily until discharge

SECONDARY OUTCOMES:
Requirements for pain medications; complications | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada